CLINICAL TRIAL: NCT04218487
Title: The Efficacy and Safety of Xuefu Zhuyu Capsule in Treating "Qizhi Xueyu Zheng" (Qi Stagnation and Blood Stasis Syndrome): a Randomized, Double-blind, Placebo-controlled, Adaptive Enrichment, Multicenter Controlled Trial
Brief Title: Xuefu-Zhuyu Capsule for the Treatment of "Qizhi Xueyu Zheng" (Qi Stagnation and Blood Stasis Syndrome)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhong Wang (Other)
Responsible Party: Sponsor-Investigator, Zhong Wang, Professor, China Academy of Chinese Medical Sciences
Organization: China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XFZY-V3.0
Record Dates: First submitted 2019-12-29; First posted 2020-01-06 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Chinese Medicine; Stable Coronary Heart Disease; Chronic Insomnia; Headache; Endometriosis
Keywords: Adaptive design; Qizhi Xueyu Zheng; Enrichment design
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Headache; Endometriosis | interventions — Xue-Fu-Zhu-Yu decoction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XFZY group (Experimental): 2.4g (6 capsules) three times daily for 12 weeks
  Interventions: Drug: Xuefu-Zhuyu Capsule; Other: conventional therapy
- Control group (Placebo Comparator): 2.4g (6 capsules) three times daily for 12 weeks
  Interventions: Drug: placebo; Other: conventional therapy

INTERVENTIONS:
Drug: Xuefu-Zhuyu Capsule — treatment with 2.4g (6 capsules) of XFZY three times daily for 12 weeks.
  Arms: XFZY group
Drug: placebo — treatment with 2.4g (6 capsules) of placebo three times daily for 12 weeks.
  Arms: Control group
Other: conventional therapy — conventional therapy will be given according to the suffering diseases including stable coronary heart disease, chronic insomnia, headache, endometriosis.

SUMMARY:
"Xuefu-Zhuyu capsule" (XFZY) is made from a classic Fangji "Xuefu-Zhuyu Decoction" in an ancient Chinese medical book "Yi Lin Gai Cuo" by Chinese physician Wang Qingren, which is the most representative formula for the treatment of "Qizhi-Xueyu Zheng" (Qi Stagnation and Blood Stasis Syndrome). XFZY concludes 11 kinds of Chinese herbs: Danggui(Angelica sinensis), Honghua(Safflower Flower), Chishao(Paeoniae Radix Rubra), Shengdihuang(Radix Rehmanniae), Taoren(Peach Seed), Zhike(Fructus Aurantii), Jugeng(Platycodon grandiflorum), Chuanxiong(Rhizome of Chuanxiong), Chaihu(Radix Bupleuri), Chuanniuxi(Cyathula Officinalis),Gancao(liquorice).It is mainly used to treat "Qizhi-Xueyu Zheng", which includes the symptoms such as different types of pain, irritability or depression, insomnia, chest tightness, dark skin, lumps or masses in vitro or in vivo, petechiae on the tongue, and dark purple tongue. The purpose of the trial is to evaluate the efficacy and safety of XFZY in treating "Qizhi-Xueyu Zheng", and investigate the most suitable diseases of XFZY.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria of "Qizhi Xueyu Zheng" (Qi Stagnation and Blood Stasis Syndrome).
* Meet the diagnostic criteria of stable coronary heart disease, chronic insomnia, headache (Migraine without Aura and Tension-Type Headache ), or endometriosis, among which:

  * the score of angina pectoris frequency domain in SAQ ≤ 80 points in the patients with stable coronary heart disease;
  * Pittsburgh sleep quality index> 10 points in patients with chronic insomnia;
  * Patients with migraine without aura have 3 or more attacks per month within 3 months before enrollment;
  * In patients with tension-Type headache, within 3 months before enrollment, the number of attack days per month is ≥ 2 days;
  * The VAS score of the pain ≥ 40 points in patients with endometriosis;
  * Patients with endometriosis diagnosed with any type of confirmed pathological reports(previous diagnosis is also possible).
* Patients were ≥18 and ≤75 years of age.
* Voluntarily provided written informed consent.

Exclusion Criteria:

* Patients with acute myocardial infarction, rapid atrial fibrillation, atrial flutter, paroxysmal ventricular tachycardia and other severe arrhythmias and severe cardiac and pulmonary insufficiency in the past 3 months
* Patients with acute cerebrovascular disease such as cerebral infarction and cerebral hemorrhage in the past 3 months;
* Those with poorly controlled hypertension (systolic blood pressure ≥160mmHg or diastolic blood pressure ≥100mmHg after treatment);
* Patients with aortic dissection;
* Patients with abnormal liver and kidney function indicators (ALT, AST are 1.5 times greater than the upper limit of normal value, and Scr is greater than the upper limit of normal value);
* SAS≥70 points;
* SDS≥73 points;
* VAS≥80 points;
* Patients with severe primary heart, brain, liver, kidney, and hematopoietic diseases;
* Women during pregnancy and lactation;
* Those with cognitive impairment, consciousness impairment or mental illness, who cannot communicate normally;
* People with allergies, or those who are known to be allergic to the trial drug (including its components);
* Surgery(including intervention, radio frequency, etc.) during the past 4 weeks;
* Those with bleeding tendency;
* Those who suspect or have a history of alcohol or drug abuse;
* Participation in another trial in the past 1 month;
* Other circumstances judged by the researcher to be unsuitable for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2019-12-31 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline the Chinese Medicine patient-reported-outcome scale in patients with Qizhi-Xueyu-Zheng (Qizhi-Xueyu-Zheng PRO Scale) | at 12 Week
  The Qizhi-Xueyu-Zheng PRO Scale is uesd to access the quality of life on the physical and mental health for the patients with Qizhi Xueyu Zheng. The higher score of this PRO scale indicates higher quality of life. Compared with the baseline, if the improvement of the PRO sacle is more than 30% after treatment, it indicates the effectiveness of the drug.
  s

SECONDARY OUTCOMES:
The single symptom and sign scale of Qizhi Xueyu Zheng | Baseline，4，8，12 Week
  According to the degree of symptoms and signs, the score will be assigned as follows: no = 0; mild = 1; moderate = 2; or severe = 3.
The pain scale Qizhi Xueyu Zheng | Baseline，4，8，12 Week
  The total score includes a visual analogue scale pain index and the score of degree, duration, and frequency of pain. The location of the pain will be recorded independently. The total score ranges from 0 to 19, higher score indicating severer pain.
Self-rating anxiety scale (SAS) | Baseline，4，8，12 Week
  The SAS scale consists of 20 items each which were scored from 1 to 4. The final score was calculated as the summation of all of the items which was then multiplied by a factor of 1.25. The score ranged from 50-59 indicates mild anxiety；The score from 60-69 indicates moderate anxiety；The score from 60-69 indicates severe anxiety.
Self-rating depression scale (SDS) | Baseline，4，8，12 Week
  The SDS scale consists of 20 items each which were scored from 1 to 4. The final score was calculated as the summation of all of the items which was then multiplied by a factor of 1.25. The score ranged from 50-59 indicates mild depression；The score from 60-69 indicates moderate depression；The score from 60-69 indicates severe depression.
SF-36 Quality of Life Scale | Baseline，4，8，12 Week
  SF-36 Quality of Life Scale is used to assess the health-related quality of life of patients, which is a multi-purpose, short-form health survey with 36 items. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary scores and a preference-based health utility index. The SF-36 consists of items: assessing physical functioning (PF-10 items),social functioning (SF-2 items), role limitation due to physical health (RP-4 items),bodily pain (BP-2 items),mental health (MH-5 items),role limitations due to emotional health (RE-3 items),vitality (VT-4 items);general health perceptions (GH-5 items);reported health transition (1 item).
Level of the 5-hydroxytryptamine(5-HT) | Baseline，4，8，12 Week
Level of the high-sensitivity C-reactive protein | Baseline，4，8，12 Week

OTHER OUTCOMES:
The changes of the expression files on the RNA level via the RNA sequencing in 120 patients | Baseline，4，8，12 Week
  Using the nested case-control study，60 patients with effective effect and the paired 60 patients in the control group will be taken with RNA sequencing.
The changes of the expression files on the protein level via the quantitative proteomics in 120 patients | Baseline，4，8，12 Week
  Using the nested case-control study，60 patients with effective effect and the paired 60 patients in the control group will be taken with quantitative proteomics.
The changes of Metabolomics profile in 120 patients | Baseline，4，8，12 Week
  Using the nested case-control study，60 patients with effective effect and the paired 60 patients in the control group will be taken with metabolomics.

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Wang, M.D., Study Director — Institute of Basic Chinese Medical Sciences, China Academy of Chinese Medical Sciences; Qing-Quan Liu, Prof., Principal Investigator — Beijing Hospital of Traditional Chinese Medicine
Locations (12):
- China (12):
  - Anqing Municipal Hospital, Anqing, Anhui
  - Beijing Hospital of Traditional Chinese Medicine, Capital Medical University, Beijing, Beijing Municipality
  - Dongfang Hospital of Beijing University of Chinese Medicine, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - Luohe Hospital of Chinese Medicine, Luohe, Henan
  - Nanyang Traditional Chinese Medicine Hospital, Nanyang, Henan
  - Wuhan Puren Hospital, Wuhan, Hubei
  - Taizhou Second People's Hospital, Taizhou, Jiangsu
  - Liaoyuan Hospital of Traditional Chinese Medicine, Liaoyuan, Jilin
  - Affiliated Hospital of Inner Mongolia University for the Nationalities, Tongliao, Neimenggu
  - First Teaching Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality